CLINICAL TRIAL: NCT00139451
Title: Nutrients and Hormones: Effects in Boys With Disordered Growth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Nelly Mauras, Chief, Division of Endocrinology, Diabetes & Metabolism, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 04-016
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Constitutional Growth Delay; Nutrition Disorders; Growth Disorders
Keywords: GH; Delayed Growth; Energy Expenditure; Puberty; Nutrition; Short Stature
MeSH Terms: conditions — Puberty, Delayed; Nutrition Disorders; Growth Disorders; Dwarfism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition and Growth Hormone (Active Comparator)
  Interventions: Drug: Pediasure; Drug: GH
- Observation and Growth Hormone (Active Comparator)
  Interventions: Drug: GH

INTERVENTIONS:
Drug: Pediasure — With the assistance of a research dietician, we will prescribe and monitor the use of a liquid food supplement (Pediasure). Adjustments to the supplementation will be made based on weight measurements in the clinic with subjects wearing paper gowns at 2 and 4w, and monthly thereafter, and repeat dietary intake and TEE assessment at 6 and 12mo.
  Arms: Nutrition and Growth Hormone
Drug: GH — Growth Hormone will be 0.3mg/kg/week, given SC once daily.

SUMMARY:
The purpose of the study is to find out if patients with constitutional delay of growth have a mismatch between energy intake and utilization (as measured by doubly labeled water) and to compare the improvement in growth and energy balance between a group of boys treated with growth hormone (GH) alone versus those given GH plus added nutritional supplements for one year.

DETAILED DESCRIPTION:
Two groups of boys 7-10 years old who are very short and below average in weight but otherwise healthy will be studied. One group will be observed initially for 6 months and then receive GH injections every day for the subsequent 12 months. Another group of boys will get a high-calorie drink every day for 6 months, and then receive GH injections plus the supplement every day for the next 12 months. We will compare how well boys grow in height, weight and the changes in body composition. We will compare diet and energy usage using the doubly labeled water technique. A battery of hormonal and nutritional tests will be performed, as well as body composition assessment.

ELIGIBILITY:
Inclusion Criteria:

* Boys 7-10 years old who are very short and below average in weight but otherwise healthy.
* Delay in skeletal maturation > 1 year.

Exclusion Criteria:

* Growth hormone deficiency
* Chronic illness
* Participation in high endurance athletics

Ages: 7 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2004-05; Primary Completion 2007-12 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in height, weight, and body composition | 6month, 12month, 18month

SECONDARY OUTCOMES:
Changes in total energy expenditure | 6month, 12month

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mauras, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- See also: issues related to child health — http://kidshealth.org